CLINICAL TRIAL: NCT00312000
Title: A Randomised Study of Sequential Versus Combination Chemotherapy in Patients With Previously Untreated Advanced Colorectal Carcinoma
Brief Title: Sequential Versus Combination Chemotherapy in Advanced Colorectal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: Koningin Wilhelmina Fonds (Other); Sanofi (Industry); Hoffmann-La Roche (Industry)
Responsible Party: C.J.A. Punt, MD PhD, DCCG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIRO1
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Advanced Colorectal Cancer
Keywords: colorectal; cancer; capecitabine; irinotecan; oxaliplatin
MeSH Terms: conditions — Neoplasms | interventions — capecitabine-irinotecan combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1Capecitabine-irinotecan (Active Comparator): 1st line- 2nd line (3rd line oxaliplatin plus capecitabine)
  Interventions: Drug: capecitabine-irinotecan
- 2capecitabine plus irinotecan (Experimental): 1st line (2nd line oxaliplatin plus capecitabine)
  Interventions: Drug: capecitabine+irinotecan (1st line)

INTERVENTIONS:
Drug: capecitabine-irinotecan — 1. st line capecitabine 1250 mg/m2 orally b.i.d. on day 1-14
  2. nd line q 3 w irinotecan 350 mg/m2 IV infusion on day 1
  Arms: 1Capecitabine-irinotecan
Drug: capecitabine+irinotecan (1st line) — q 3 w irinotecan 250 mg/m2 IV infusion in 30 minutes on day 1 2 hours after discontinuation of the infusion followed by capecitabine 1000 mg/m2 orally b.i.d. on day 1-14
  Arms: 2capecitabine plus irinotecan

SUMMARY:
Primary objective:To assess the efficacy, defined as overall survival, of sequential versus combination chemotherapy for advanced colorectal cancer (CRC).

Methodology Open, randomised multicenter phase III study. Randomisation by centre will be centralized. 820 patiënts with histologically proven advanced CRC; not amenable to curative surgery. Measurable or evaluable disease. Age 18 years and above. WHO performance status 0-2.

Test products:

Arm A: First line: capecitabine capecitabine 1250 mg/m2 orally b.i.d. on day 1-14 (q3),until progression or unacceptable toxicity. Second line: irinotecan 350 mg/m2 IV infusion on day 1 (q3),until progression or unacceptable toxicity. Third line: oxaliplatin 130 mg/m2 IV infusion on day 1 and capecitabine 1000 mg/m2 orally b.i.d. on day 1-14 (q3). Arm B: First line: irinotecan 250 mg/m2 IV infusion in 30 minutes on day 1 and capecitabine 1000 mg/m2 orally b.i.d. on day 1-14 (q3), until progression or unacceptable toxicity. Second line: oxaliplatin 130 mg/m2 IV on day 1 and capecitabine 1000 mg/m2 orally b.i.d. on day 1-14 (q3), until progression or unacceptable toxicity.

Patients will be followed by CT-scan every 9 weeks for response while on treatment, or at any other moment when progression is suspected. After cessation of chemotherapy, patients will be followed every 3 months until death. Clinical and laboratory toxicity/symptomatology will be graded according to NCI common criteria.

DETAILED DESCRIPTION:
Objectives: Primary objective:

To assess the efficacy, defined as overall survival, of sequential versus combination chemotherapy for advanced CRC.

Secondary objectives are to assess:

To assess Tumour response (CR, PR or SD) Progression free survival Quality of life Toxicity profile Methodology Open, randomised multicenter phase III study. Randomisation by centre will be centralized by IKC. Number of patients 820 Main criteria for inclusion Histology and staging disease

* Histologically proven advanced CRC; not amenable to curative surgery;
* Of Note: In case of a single metastasis, histological or cytological proof of colorectal carcinoma should be obtained prior to randomisation.
* Measurable or evaluable disease. Serum CEA as the only parameter for disease activity is not allowed.

General conditions

* Written informed consent;
* Age 18 years and above;
* WHO performance status 0-2;
* Adequate bone marrow function (WBC > 3.0 x 109/L, platelets > 100 x 109/L, Hb > 6 mmol/L);
* Adequate hepatic function: total bilirubin < 1. 5 x upper normal limit, ASAT and ALAT < 3 x upper normal limits (in case of liver metastases < 5 x upper normal limits);
* Adequate renal function: creatinin < 1. 5 x upper normal limits. Other
* Expected adequacy of follow-up.

Main criteria for exclusion General conditions

* Pregnancy or lactation;
* Patients (M/F) with reproductive potential not implementing adequate contraceptives measures.

Prior or current history

* Prior chemotherapy for advanced disease; prior adjuvant chemotherapy is allowed, provided that the last drug administration took place more than 6 months prior to randomisation.
* Serious concomitant diseases preventing the safe administration of chemotherapy or likely to interfere with the study assessments;
* Serious active infections;
* Inflammatory bowel disease or other diseases associated with chronic diarrhoea;
* Previous extensive irradiation of pelvis or abdomen;
* Other malignancies in the past 5 years with the exception of adequately treated carcinoma in situ of the cervix or squamous or basal cell carcinoma of the skin.

Concomitant treatments

* Concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation;
* Concurrent treatment with any other anti-cancer therapy. Test product, dose and mode of administration Arm A First line: capecitabine

Every 3 weeks (q 3):

capecitabine 1250 mg/m2 orally b.i.d. on day 1-14. This schedule will be continued until progression or unacceptable toxicity. Continuation after 6 months without disease progression and/or severe toxicity at the investigator's discretion.

Second line: irinotecan

Every 3 weeks (q 3):

irinotecan 350 mg/m2 IV infusion on day 1. This schedule will be continued until progression or unacceptable toxicity. Continuation after 6 months without disease progression and/or severe toxicity at the investigator's discretion.

Third line: oxaliplatin plus capecitabine oxaliplatin 130 mg/m2 IV infusion on day 1 and capecitabine 1000 mg/m2 orally b.i.d. on day 1-14. This schedule will be continued until progression or unacceptable toxicity. Continuation after 6 months without disease progression and/or severe toxicity at the investigator's discretion.

Arm B First line: irinotecan plus capecitabine

Every 3 weeks (q 3):

irinotecan 250 mg/m2 IV infusion in 30 minutes on day 1 2 hours after discontinuation of the infusion followed by capecitabine 1000 mg/m2 orally b.i.d. on day 1-14. This schedule will be continued until progression or unacceptable toxicity. Continuation after 6 months without disease progression and/or severe toxicity at the investigator's discretion.

Second line: oxaliplatin plus capecitabine

Every 3 weeks (q 3):

oxaliplatin 130 mg/m2 IV infusion in 2 hours on day 1 and capecitabine 1000 mg/m2 orally b.i.d. on day 1-14. This schedule will be continued until progression or unacceptable toxicity. Continuation after 6 months without disease progression and/or severe toxicity at the investigator's discretion.

Duration of treatment and follow-up Treatment is continued until disease progression, or unacceptable toxicity. Patients will be followed by CT-scan every 9 weeks for response while on treatment, or at any other moment when progression is suspected. After cessation of chemotherapy, patients will be followed every 3 months until death. Death or progression should be reported whenever it occurs.

Criteria for evaluation Efficacy All patients will be included in the survival analysis (intent-to-treat). All patients receiving > 9 weeks of treatment (i.e. 3 cycles) will be considered evaluable for response, unless documented progression occurred earlier.

Safety profile Safety will be analysed in each treatment group. Patients having received > treatment doses are evaluable for toxicity. Evaluation will be performed by patient and by cycle on the intent-to-treat population. Clinical and laboratory toxicity/symptomatology will be graded according to NCI common criteria. The adverse events which are not reported in NCI common criteria will be graded as: mild, moderate, severe, life threatening.

Statistical methodology The expected median survival in Arm A (standard arm) is 14 months. It is anticipated that the median survival in Arm B (experimental arm) will be 19 months. 620 patients (310 in each arm) are needed to show this increase in median survival (>=0,05 and >=0,80).

Stratification parameters Patients will be stratified for the following parameters:

* WHO performance status 0-1 vs 2
* Serum LDH normal versus above normal
* Prior adjuvant therapy versus no prior adjuvant therapy
* Predominant localisation of metastases in the liver vs extrahepatic site(s)
* Per participating institution

ELIGIBILITY:
Inclusion Criteria:

* Histology and staging disease

  * Histologically proven CRC; advanced disease, not amenable to curative surgery;
  * Of Note: In case of a single metastasis, histological or cytological proof of colorectal carcinoma should be obtained prior to randomisation.
  * Measurable or evaluable disease; Serum CEA as the only parameter for disease activity is not allowed.
* General conditions

  * Written informed consent;
  * Age 18 years and above;
  * WHO performance status 0-2;
  * Adequate bone marrow function(WBC > 3.0 x 109/L, platelets > 100 x 109/L, Hb > 6 mmol/L);
  * Adequate hepatic function: total bilirubin < 1. 5 x upper normal limit, ASAT and ALAT < 3 x upper normal limits; in case of liver metastases < 5 x upper normal limits
  * Adequate renal function: creatinin < 1. 5 x upper normal limits.
* Other - Expected adequacy of follow-up.

Exclusion Criteria:

* General conditions

  * Pregnancy or lactation;
  * Patients (M/F) with reproductive potential not implementing adequate contraceptives measures.
* Prior or current history

  * Prior chemotherapy for advanced disease; prior adjuvant chemotherapy is allowed provided that the last administration was given > 6 months prior to randomisation.
  * Serious concomitant diseases preventing the safe administration of chemotherapy or likely to interfere with the study assessments;
  * Serious active infections;
  * Inflammatory bowel disease or other diseases associated with chronic diarrhoea;
  * Previous extensive irradiation of the pelvis or abdomen;
  * Other malignancies in the past 5 years with the exception of adequately treated carcinoma in situ of the cervix or squamous or basal cell carcinoma of the skin.
* Concomitant treatments

  * Concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation;
  * Concurrent treatment with any other anti-cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2003-01; Primary Completion 2006-02 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | study duration

SECONDARY OUTCOMES:
Tumour response | study duration
Progression free survival | study duration
Quality of life | study duration
Toxicity profile | study duration

CONTACTS AND LOCATIONS:
Overall Officials: C. J. A. Punt, Prof.Dr., Principal Investigator — University Medical Center St. Radboud, Nijmegen, The Netherlands

REFERENCES:
- [Result] Koopman M, Antonini NF, Douma J, Wals J, Honkoop AH, Erdkamp FL, de Jong RS, Rodenburg CJ, Vreugdenhil G, Akkermans-Vogelaar JM, Punt CJ. Randomised study of sequential versus combination chemotherapy with capecitabine, irinotecan and oxaliplatin in advanced colorectal cancer, an interim safety analysis. A Dutch Colorectal Cancer Group (DCCG) phase III study. Ann Oncol. 2006 Oct;17(10):1523-8. doi: 10.1093/annonc/mdl179. Epub 2006 Jul 27. PMID 16873425
- [Result] Koopman M, Antonini NF, Douma J, Wals J, Honkoop AH, Erdkamp FL, de Jong RS, Rodenburg CJ, Vreugdenhil G, Loosveld OJ, van Bochove A, Sinnige HA, Creemers GM, Tesselaar ME, Slee PHTJ, Werter MJ, Mol L, Dalesio O, Punt CJ. Sequential versus combination chemotherapy with capecitabine, irinotecan, and oxaliplatin in advanced colorectal cancer (CAIRO): a phase III randomised controlled trial. Lancet. 2007 Jul 14;370(9582):135-142. doi: 10.1016/S0140-6736(07)61086-1. PMID 17630036
- [Derived] van Kessel CS, Samim M, Koopman M, van den Bosch MA, Borel Rinkes IH, Punt CJ, van Hillegersberg R. Radiological heterogeneity in response to chemotherapy is associated with poor survival in patients with colorectal liver metastases. Eur J Cancer. 2013 Jul;49(11):2486-93. doi: 10.1016/j.ejca.2013.03.027. Epub 2013 May 18. PMID 23692811
- See also: site of the Dutch Colorectal Cancer Group — http://www.dccg.nl